CLINICAL TRIAL: NCT05867108
Title: Contribution of the Sonication of Implants to the Diagnosis of Joint Prosthesis Infection: Retrospective Cohort Study From 2019 to 2022 at the University Hospitals of Strasbourg
Brief Title: Contribution of the Sonication of Implants to the Diagnosis of Joint Prosthesis Infection: A Retrospective Cohort Study
Acronym: SonicHUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8956
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-05

CONDITIONS: Prosthesis Related Infection
Keywords: Prosthesis Related Infection; Joint prosthesis infection; Sonication of implants; Cutibacterium acnes; Streptococci
MeSH Terms: conditions — Prosthesis-Related Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Studies on sonication suffer from a heterogeneity which makes their analysis complex, due to the absence of a gold standard allowing positive cases to be defined unequivocally. Thus, the sensitivity of the technique has been assessed on cases defined in different ways, which makes the studies difficult to compare (number of samples taken, number of positive samples, variable duration of culture, etc.). It should nevertheless be noted that the majority of the series conclude with a higher sensitivity than that of standard samples, in particular in the event of a strain with difficult growth (Cutibacterium acnes, deficient Streptococci) or in the event of prior antibiotic therapy.

In the absence of a comparative reference allowing to conclude on the intrinsic performances of sonication as a diagnostic test, it seems interesting to evaluate its contribution in current practice, in particular in the difficult cases where the standard culture does not make it possible to fulfill the criterion. major (zero or only one positive sample). To the knowledge of the investigators, there is no study of this kind, which could make it possible to specify the place of this technique in the diagnostic procedure and to improve the care of patients.

ELIGIBILITY:
Inclusion criteria:

* Adult patients (age ≥18 years)
* Have been hospitalized and operated on for a change of hip or knee joint prosthesis between 01/01/2019 and 07/31/2022
* Have had at least 3 samples taken for microbiological purposes, pre- or intraoperatively
* the explanted prosthesis must have been analyzed by sonication.
* not opposing the reuse of its data for scientific research purposes

Exclusion criteria:

- Opposition of the patient to the reuse of his data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (age ≥18 years) have been hospitalized and operated on for a change of hip or knee joint prosthesis between 01/01/2019 and 07/31/2022
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-03 (Estimated); Study Completion 2024-03-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with only a peri-prosthetic sample whose culture is positive, and for whom the culture of the sonication fluid is positive and consistent with this first sample, with an objective of >5%. | 4 years after implant

CONTACTS AND LOCATIONS:
Overall Officials: Cécile RONDE-OUSTAU, MD, Study Director — University Hospitals of Strasbourg
Locations (1):
- ervice de Chirurgie Orthopédique Septique - CHU de Strasbourg - France, Strasbourg, France